CLINICAL TRIAL: NCT07045350
Title: Evaluation of the Effects of Dexamethasone-Enriched Platelet-Rich Fibrin on Postoperative Pain, Edema, and Trismus Following Impacted Mandibular Third Molar Surgery: A Randomized Split-Mouth Clinical Trial
Brief Title: Dexamethasone-PRF in Mandibular Third Molar Surgery: Effect on Pain, Edema, and Trismus (DEXPRF-3M)
Acronym: DEXPRF-3M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Muhammet Caner Dere, PhD, Cumhuriyet University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCU-EC-No: 2023-07/02; DIS-2024-328 (Other Grant/Funding Number: CÜBAP, Sivas Cumhuriyet University)
Record Dates: First submitted 2025-06-18; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Impacted Mandibular Third Molar
Keywords: Third molar; Platelet Rich Fibrin; Dexamethasone; Edema; Pain; Trismus
MeSH Terms: conditions — Edema; Pain; Trismus

STUDY DESIGN:
Intervention Model Description: This randomized controlled clinical trial uses a split-mouth design, where each patient serves as their own control. One side receives platelet-rich fibrin (PRF) from dexamethasone-enriched blood, while the contralateral side receives standard PRF to compare postoperative outcomes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and clinicians performing postoperative evaluations were blinded to the treatment allocation. This was done to minimize bias in reporting and assessment of postoperative pain, edema, and trismus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard PRF (Active Comparator): Application of standard platelet-rich fibrin (PRF) prepared from blood without dexamethasone to the mandibular third molar extraction site.
  Interventions: Procedure: Platelet-rich fibrin (PRF)
- Test - Dexamethasone-enriched PRF (Experimental): Application of platelet-rich fibrin (PRF) prepared from blood enriched with 4 mg dexamethasone to the mandibular third molar extraction site.
  Interventions: Procedure: Platelet-rich fibrin (PRF)

INTERVENTIONS:
Procedure: Platelet-rich fibrin (PRF) — Application of autologous platelet-rich fibrin (PRF) prepared from peripheral blood with or without the addition of 4 mg dexamethasone directly into the blood collection tube prior to centrifugation. PRF was applied into the extraction socket after impacted mandibular third molar surgery. The test group received PRF prepared from blood enriched with dexamethasone, while the control group received standard PRF without dexamethasone, to evaluate postoperative pain, edema, and trismus.
  Other Names: Dexamethasone-Enriched Platelet-Rich Fibrin

SUMMARY:
Brief Summary

This clinical trial investigates the effects of platelet-rich fibrin (PRF) derived from dexamethasone-enriched blood on postoperative recovery following the surgical extraction of impacted mandibular third molars (wisdom teeth). The study aims to determine whether the addition of dexamethasone, a potent anti-inflammatory medication, to the blood used for PRF preparation can reduce postoperative pain, swelling, and limited mouth opening (trismus) more effectively than standard PRF.

The study is designed as a randomized, split-mouth, double-blind clinical trial involving 16 patients who require bilateral extraction of impacted lower third molars. Each patient receives both treatments: one extraction socket treated with standard PRF and the other with dexamethasone-enriched PRF. Postoperative outcomes including pain intensity, edema, trismus, and analgesic consumption are recorded and analyzed.

The results of this study could offer a safer and more effective method for managing discomfort after wisdom tooth removal, potentially improving patient quality of life and reducing the need for additional medications.

DETAILED DESCRIPTION:
Detailed Description

Background:

Third molar (wisdom tooth) extraction is a common oral surgical procedure often associated with postoperative inflammatory complications such as pain, edema, and trismus, which can significantly reduce patient quality of life. Platelet-rich fibrin (PRF) has been used to enhance healing and reduce postoperative morbidity. Dexamethasone is a corticosteroid known for its potent anti-inflammatory effects. This study evaluates whether PRF prepared from dexamethasone-enriched blood can improve postoperative outcomes compared to standard PRF.

Objectives:

The primary objective is to assess the effect of dexamethasone-enriched PRF on postoperative pain following impacted mandibular third molar extraction. Secondary objectives include evaluation of edema, trismus, and analgesic consumption.

Study Design:

This is a randomized, controlled, split-mouth, double-blind clinical trial conducted in a single center. Sixteen patients with bilateral symmetrical impacted mandibular third molars requiring extraction were enrolled. Each patient received two different treatments: one socket treated with standard PRF and the contralateral socket treated with dexamethasone-enriched PRF.

Participants:

Eligible patients were aged 18-25 years, in good systemic health, with no contraindications for oral surgery or corticosteroid use. Exclusion criteria included systemic diseases, pregnancy or lactation, hypersensitivity to corticosteroids, poor oral hygiene, recent corticosteroid therapy, and temporomandibular joint disorders.

Intervention:

Peripheral venous blood was drawn from each patient, with dexamethasone added to one sample prior to centrifugation to prepare the test PRF. The control PRF was prepared without dexamethasone. PRF clots were applied immediately into the extraction sockets after tooth removal.

Outcome Measures:

Postoperative pain was measured using a visual analog scale (VAS) at 24, 48, and 72 hours. Edema and trismus were evaluated on postoperative days 1, 3, and 7. Analgesic intake was recorded throughout the postoperative period. Data were analyzed with appropriate statistical tests considering p < 0.05 as significant.

Ethical Considerations:

The study was approved by the institutional ethics committee (approval number XXXX), and written informed consent was obtained from all participants. The study complied with the Declaration of Helsinki guidelines.

Significance:

Findings from this study may provide evidence for a novel, autologous drug delivery method to reduce postoperative morbidity after mandibular third molar surgery, potentially improving patient comfort and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 25 years.
* Presence of bilateral, symmetrical, bone-retained impacted mandibular third molars requiring extraction.
* Systemically healthy individuals with no chronic medical conditions.
* Good oral hygiene and healthy periodontal status.
* Radiographically confirmed bilateral similarity of impacted third molars.
* Patients willing to participate and who provided written informed consent.

Exclusion Criteria:

* Presence of systemic diseases or conditions that may affect wound healing.
* Regular use of prescription medications.
* Pregnant or lactating individuals, or those with suspected pregnancy.
* Known allergy or hypersensitivity to dexamethasone or related compounds.
* Poor oral hygiene or active periodontal disease.
* Presence of fungal, viral, or bacterial infection either systemically or locally.
* History of corticosteroid use within the past month.
* Temporomandibular joint disorders affecting mouth opening.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain and Analgesic Consumption | 72 hours post-surgery
  Measurement of postoperative pain using the Visual Analog Scale (VAS; range 0-10, where 0 indicates no pain and 10 indicates the worst imaginable pain) and total analgesic intake at 24, 48, and 72 hours after mandibular third molar extraction.

SECONDARY OUTCOMES:
Postoperative Facial Edema | Postoperative days 1, 3, and 7
  Facial swelling will be evaluated by measuring linear distances between predefined facial landmarks (tragus-commissure, tragus-pogonion, lateral canthus-gonion) on postoperative days 1, 3, and 7.
Postoperative Trismus | Postoperative days 1, 3, and 7
  Maximum interincisal mouth opening (in millimeters) will be measured preoperatively and on postoperative days 1, 3, and 7 using a digital caliper to assess trismus severity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Caner Dere, DDS, Principal Investigator — Sivas Cumhuriyet University, Faculty of Dentistry
Locations (1):
- Sivas Cumhuriyet University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be available upon request from the corresponding author (Dr. Muhammet Caner Dere, caner_1995@hotmail.com). The shared data will include anonymized individual participant data related to postoperative pain, edema, trismus, and analgesic use. Data will be available after study completion and publication, for a period of 5 years. The data will be shared for scientific research and meta-analyses, subject to ethics committee approval and a data use agreement. Participants' informed consent included agreement for anonymized data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The individual participant data (IPD) and supporting materials will be available from 6 months after publication of the final results and for a period of 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal will be granted access to anonymized individual participant data (IPD), including postoperative pain scores, edema, trismus measurements, and analgesic intake. Access will be provided for the purpose of scientific research or meta-analyses, subject to approval by an ethics committee and after signing a data use agreement. Data will be available by contacting the corresponding author.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT07045350/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT07045350/ICF_001.pdf